CLINICAL TRIAL: NCT02517593
Title: Genetic Risk Estimation of Breast Cancer Prior to Preventive Medication Uptake: A Pilot Study to Determine if a Polygenic Risk Score Influences the Decision to Accept Breast Cancer Preventive Medications (Tamoxifen, Raloxifene, or Exemestane) Amongst Non-BRCA Women at Risk
Brief Title: Genetic Risk Estimation of Breast Cancer Prior to Preventive Medication Uptake
Acronym: GENRE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Sandhya Pruthi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-006204; CCM-003 (Other: CancerCare Manitoba)
Record Dates: First submitted 2015-07-31; First posted 2015-08-07 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: BCRAT; IBIS; PRS; breast cancer; Tyrer-Cuzick
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRS (Other): Providing polygenic risk score (PRS)
  Interventions: Genetic: Polygenic Risk Score

INTERVENTIONS:
Genetic: Polygenic Risk Score — A Polygenic Risk Score (PRS) is a blood based genetic test which assesses 77 common breast cancer susceptibility loci (Single Nucleotide Polymorphisms). The PRS has been retrospectively validated and categorizes women into three categories of lifetime risk of developing breast cancer: Low Risk (<15% lifetime risk), Above Average Risk (15 to 40%), and high risk (>40%).
  Other Names: PRS

SUMMARY:
The primary aim of this study is to determine if the addition of an individual polygenic risk score (PRS), in addition to the standard National Cancer Institute's Breast Cancer Risk Assessment Tool (BCRAT) or Tyrer-Cuzick (IBIS) score, will aid women at risk of breast cancer in making a decision to take (or not take) medications to prevent breast cancer

DETAILED DESCRIPTION:
This trial is a prospective pilot study looking to integrate a novel and retrospectively validated polygenic risk score (PRS), based on 77 Single Nucleotide Polymorphisms (SNPs), into a standard breast cancer prevention consultation for non-BRCA women. In order to be eligible for trial participation, women will need to have a BCRAT estimate of ≥3% for the 5 year risk of developing breast cancer (which corresponds to the United States Preventative Services Task Force threshold for moderate to strong benefit from breast cancer preventing medications such as tamoxifen or raloxifene.

At the time of the breast cancer prevention consultation, women will be offered participation in this study by a clinical trials nurse and informed written consent will be obtained. For consenting patients, a single 7 to 10 ml blood sample will be taken and couriered to the MAYO clinic for sample analysis and several surveys will be administered. One of the surveys will assess the participants understanding and intention to take or not take breast cancer preventing medications. The decision to take or not take a breast cancer preventing medication will be deferred until a subsequent follow up visit.

On the second visit, the PRS test results will be reviewed with the patient and a recommendation regarding preventive medications will be made. The PRS score will risk stratify patients into one of three lifetime risk categories of developing breast cancer (low risk (<15 % lifetime risk), above average risk (15 to <40% risk) and high risk (>40%)). Participants will then answer a second survey in which their understanding of their breast cancer risk and intention to take breast cancer preventing medications will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Women > 35 years old and < 75 years old
2. Women with either of the following:

   A. a NCI-BCRAT 5 year risk of ≥ 3% which corresponds to the level in which there is moderate evidence of treatment benefit outweighing risk according to the US Preventative Services Task Force (32); or B. Women with a IBIS (Tyrer-Cuzik) score for the 10 year risk of breast cancer of ≥5%
3. Able to participate in all aspects of the study
4. Understand and signed the study informed consent

Exclusion Criteria:

1. Women whose BCRAT falls below the threshold (<3 % 5 year risk) of moderate benefit according to the US Preventative Task Force AND Women whose IBIS score is <5% for the 10 year risk
2. Women with known BRCA1 and BRCA2 mutations
3. Women with known contra-indications to Tamoxifen, raloxifene or exemestane
4. Unable to give informed consent
5. Prior history of invasive breast cancer or ductal carcinoma in situ
6. At risk due to prior radiation therapy to the chest

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Patient self-reported intention to take a breast cancer preventing medication | up to 6 months after initial consultation

SECONDARY OUTCOMES:
Proportion of patients who are taking preventive medications at year 1 | 1 year
Proportion of patients who are taking preventive medications at year 2 | 2 years
Endocrine related quality of life scores at 1 year | 1 year
  Functional Assessment of Cancer Therapy (FACT) - Endocrine Subscale Quality of Life Tool
Endocrine related quality of life scores at 2 years | 2 years
  Functional Assessment of Cancer Therapy (FACT) - Endocrine Subscale Quality of Life Tool

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Pruthi, MD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials